CLINICAL TRIAL: NCT02142075
Title: Population Pharmacokinetic (PK) Study of Multiple Doses of Cubicin® (Daptomycin) 10 mg/kg in Critical Care Patients Having Bacteremia, Endocarditis or Skin Soft Tissue Infections Due to Gram Positive Bacteria With Various Degrees of Renal Failure
Acronym: DAPTOREA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DAPTOREA
Record Dates: First submitted 2014-03-12; First posted 2014-05-20 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Renal Failure; Critical Care; Gram Positive Bacteria
Keywords: Pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency | interventions — Daptomycin

ARMS (1):
- Daptomycin, IV (Experimental): * Patients with creatinine clearance ≥30 ml/min will receive 10 mg/kg of daptomycin (Cubicin®) once daily,
  * Patients with creatinine clearance <30 ml/min will receive the same daptomycin dose (10 mg/kg) but less frequently, every 48h instead of every day
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin

SUMMARY:
Treatment of infections in critically ill patients remains a significant challenge to intensivists world-wide with persisting high mortality and morbidity. Compelling evidence suggests that source control of the pathogen and appropriate antibiotic therapy remain the most important interventions to improve patients' outcome, the latter including the administration of a suitable molecule at an optimized dosage regimen.

Daptomycin is the first representative of a new family of antibiotics, the cyclic lipopeptides. Its bactericidal effect against Gram-positive bacteria, including meticillin-resistant strains, and its low renal toxicity, make it a useful antibiotic in critically ill patients having infections due to resistant Gram positive strains.

Unfortunately, no PK study has been performed in infected critically ill patients without renal replacement therapy. A vast array of pathophysiological changes can occur in infected critically ill patients, leading to changes in volume of distribution and clearance of antibiotics in these patients, which may affect the antibiotic concentration at the target site.

It is therefore important to better characterize daptomycin PK in infected patients with various degrees of renal failure in order to define optimal dosing regimens.

This project aims to identify optimal daptomycin administration schemes in critical care patients with various degrees of renal impairment

ELIGIBILITY:
Inclusion Criteria:

* Patients of two sexes aged 18 to 85 years,
* Hospitalized in one of the intensive care unit participating in the study,
* Under mechanical ventilation,
* Having skin or soft tissue infection, bacteremia or endocarditis caused by Gram positivebacteria susceptible to daptomycin,
* Having given written consent to participate to the study.
* Patients with severe sepsis and septic shock will also be included because it's the very population that may benefit from daptomycin treatment and it's important to get data for these patients in order to optimize their treatment.

Exclusion Criteria:

* Pregnant or lactating women
* Obese subjects (body mass index > 40 mg/m2)
* Patients requiring extrarenal replacement therapy,
* Patients having already received daptomycin during the 21 days prior to inclusion,
* Known hypersensitivity to daptomycin,
* History of myopathy
* creatine phosphokinase >5 upper limit of normal
* Patients not affiliated to a social security scheme,Patients deprived of their liberty by judicial or administrative decision

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2014-03; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
area under the curve / minimum inhibitory concentration ratio of distribution and elimination of daptomycin in plasma and urine | 12 months
Cmin and Cmax of distribution and elimination of daptomycin in plasma and urine | 12 months
volume of distribution of daptomycin in plasma and urine | 12 months
clearance of distribution and elimination of daptomycin in plasma and urine | 12 months

SECONDARY OUTCOMES:
the clinical and microbiological efficacy during Daptomycine treatment and two weeks after the end of it | 12 months
  Patients will be considered to have clinical failure if they will have no response to the study drug on the basis of ongoing signs and symptoms of infection. Otherwise, patients will be considered to have clinical success.
renal and muscular tolerance during Daptomycin treatment and two weeks after the end of it | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Lasocki S, University Hospital of Angers, Angers, France
  - Asehnoune K, University Hospital of Nantes, Nantes, France
  - Seguin P, University Hospital of Rennes, Rennes, France
  - Ferrandiere M, University Hospital of Tours, Tours, France